CLINICAL TRIAL: NCT01935024
Title: Assessing the Benefits of an Outpatient Aerobic Activity Program in Patients With Alzheimer's Disease
Brief Title: Benefits of Exercise in Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Carmela Tartaglia, MD, FRCPC, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-5749-AE
Record Dates: First submitted 2013-08-23; First posted 2013-09-04 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; dementia; aerobic exercise
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Activity level (No Intervention)
- Personalized Exercise Regimen (Active Comparator)
  Interventions: Other: Personalized Exercise Regimen

INTERVENTIONS:
Other: Personalized Exercise Regimen — All exercise regimens include a stationary bicycle.
  Arms: Personalized Exercise Regimen

SUMMARY:
Exercise has been shown to be beneficial for the brain. The investigators would like to test this specifically for those diagnosed with Alzheimer's disease. This study will involve 30 randomized patients to take part in the out-patient exercise program and 30 patients to continue with their regular activities over a 6-month period. Once that period is over, half of the 30 patients who participated in the outpatient exercise program will continue in the program and the other half will be randomized to independently continue to exercise. The investigators hypothesize that exercising will benefit the patient by slowing the dementia process, improving behavioral symptoms, and decreasing volume loss of certain brain regions. Each person will perform personalized exercise regimens, MR imaging and neuropsychological tests will be used to measure the benefits of exercise. Ultimately, the hope is that the results of this study could be used to facilitate exercise programs for patients. Enrollment is completely voluntary and all personal data obtained will remain confidential.

ELIGIBILITY:
Inclusion criteria for patients will be as follows:

1. Diagnosis of probable Alzheimer's disease as per 2011 criteria
2. Mild or moderate stage of dementia, a score of 10-25 in the Clinical dementia rating score (CDR) <2 and a score of 10-25 (inclusive) on the Montreal Cognitive Assessment (MoCA)
3. Age 60 to 95 inclusive
4. Mobility, preserved vision and hearing (eyeglasses and/or hearing aid are permissible) sufficient for compliance with testing procedures
5. Ability to tolerate and perform aerobic exercise program (as per The Canadian Society for Exercise Physiology; all patients above the age of 69 embarking on a new exercise routine should have the "Physical Activity Readiness Medical Examination" (PARmed-X) form completed by their family physician. All patients being asked to enroll in the study will have their PCPs fill out this form to ensure the patient is able to withstand the exercise program. If they are being followed by a cardiologist, they fill out the form)
6. Presence of a respective caregiver
7. Ability to tolerate MRI
8. Ability to speak and understand the English language (as questionnaires and tests are only available in English)

Inclusion criteria for the caregivers will be as follows:

1. Being the primary caregiver for a given patient
2. Ability to speak and understand English (as questionnaires and tests are only available in English)
3. MoCA score ≥ 26

Exclusion criteria for Patients and Caregivers:

1. History of another neurological disorder
2. Psychiatric disorder
3. Severe aphasia (semantic word loss)
4. Visual deficits requiring correction beyond the use of eyeglasses or contact lenses (intact visual acuity is required for completing both the questionnaires and the emotion evaluation test which consists of video vignettes)
5. Hearing problems requiring correction beyond hearing aids (videos have an auditory component)

Exclusion Criteria for Patients:

1. Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal pieces or objects in the eyes, skin or body will be excluded as they will be unable to have a MRI scan
2. Inability to tolerate or perform aerobic exercise as declared by family physician on PARmed-X form
3. Significant vascular disease seen on MRI (Fazekas score>2)

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-08-01 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological Test Battery | Throughout first 6 months of patient participation
  The test battery selected comprises of standardized, validated tests focusing on domains including: attention & concentration, executive functioning, learning and memory, visuospatial, language and semantic memory, pre-morbid intellectual functioning, and speed of processing.

CONTACTS AND LOCATIONS:
Overall Officials: Carmela Tartaglia, MD, FRCPC, Principal Investigator — Cognitive Neurologist at the Toronto Western Hospital Memory Clinic
Locations (1):
- Toronto Western Hospital, WW5-449, Toronto, Ontario, Canada